CLINICAL TRIAL: NCT01413334
Title: Noninvasive Diagnosis of Ischemia Causing Coronary Stenosis Using Coronary CT Angiograms (CCTA) : Comparison of Transluminal Attenuation Gradient (TAG) and Fractional Flow Reserve Computed From CCTA (FFR CT)
Brief Title: Transluminal Attenuation Gradient Versus CT Fractional Flow Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Division of cardiology/Cardiovascular center, Seoul National University Hospital
Other Study IDs: H-1106-076-366
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; CT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary computed tomographic angiography (CCTA) has emerged as a non-invasive test, accurately evaluate anatomic coronary artery stenosis. However, anatomically-obstructive coronary stenosis by CCTA demonstrates an unreliable relationship to lesion-specific ischemia. Recently, with the advance of imaging reconstruction and analysis technique, several novel parameters computed from CCTA were suggested to have added value in determining the ischemia-causing coronary stenosis. In this study, diagnostic performance of transluminal attenuation gradient (TAG) and fractional flow reserve computed form CCTA (FFR-CCTA) for the presence of hemodynamically-significant coronary stenosis, as determined by fractional flow reserve (FFR).

DETAILED DESCRIPTION:
Angiographically obtained fractional flow reserve (FFR) is a useful physiologic test for assessment of lesion-specific ischemia, and a valuable adjunct to anatomic assessment of coronary artery disease (CAD) as determined by invasive coronary angiography. However, the invasiveness and measuring difficulty of FFR make it unfamiliar to perform. Coronary computed tomographic angiography (CCTA) has emerged as a non-invasive test, accurately evaluate anatomic coronary artery stenosis. Although CCTA evaluation of CAD has been validated against invasive coronary angiography and intravascular ultrasound, anatomically-obstructive coronary stenosis by CCTA demonstrates an unreliable relationship to lesion-specific ischemia. Recently, with the advance of imaging reconstruction and analysis technique, several novel parameters computed from CCTA were suggested to have added value in determining the ischemia-causing coronary stenosis. In this study, diagnostic performance of transluminal attenuation gradient (TAG) and fractional flow reserve computed form CCTA (FFR-CCTA) for the presence of hemodynamically-significant coronary stenosis, as determined by FFR, will be compared to suggest best functional parameter noninvasively computed form CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* CCTA with >=50% stenosis in a major coronary artery (>=2.0 mm diameter)
* underwent invasive coronary angiography with FFR measurement

Exclusion Criteria:

* with CCTA of poor image quality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or known coronary artery disease (CAD) who underwent coronary CT angiography, invasive coronary angiography, and fractional flow reserve measurement between May, 2010 and January, 2011
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
fractional flow reserve | 1day
  fractional flow reserve of stenotic coronary artery

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea